CLINICAL TRIAL: NCT04194970
Title: The Effects of Monitoring Weight Bearing Protocols Following Lower Extremity Surgeries Via Mobile Application and Pressure Sensors.
Brief Title: Monitoring of Weight Bearing Protocols Via Mobile Application and Pressure Sensors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ender Ersin Avci, Research assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 09.2019.593
Record Dates: First submitted 2019-11-28; First posted 2019-12-11 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Osteochondral Lesion of Talus
Keywords: Weight bearing monitoring,; Live-biofeedback; Lower extremity; Rehabilitation; WBM smart insole system

STUDY DESIGN:
Intervention Model Description: First Step of Research: development of product that can provide live-feedback (insole with pressure sensors, mobile application) (approximately- 10 healthy volunteers) Second Step of Research: Testing this product on healthy volunteers Third Step of Research: Following up the post-operative patients with product ( Group I - monitoring with live feedback, Group II- monitoring without live-feedback) (approximately- 10 post-operative patients)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (monitoring with live-feedback system) (Experimental): WBM smart insole system is a product that can monitor the pressure under the foot and provide live feedback (if this option activated) to the user in case of exceeding the specified limits. Its components are insole with pressure sensors and mobile applications (IOS, Android). Post-operative patients (osteochondral lesion of the talus) will be monitored with the WBM smart insole system in case live feedback is turned on. We aimed to ensure the compliance of patients to specified weight bearing limits. We will follow up this grup for 6 weeks periods with WBM smart insole system. Pre-op. and post-op 6 week, we evaluate the patients in case of ankle function, pain with The American Orthopaedic Foot & Ankle Society (AOFAS) Scoring. Also we will monitor the compliance success of patients with WBM smart insole system during 6 week. The relationship with compliance to weight bearing success and AOFAS scores will be evaluate.
  Interventions: Device: With WBM smart insole system to monitor compliance of specified weight bearing limits data in live feedback on and off situations
- Group II (monitoring without live feedback) (Active Comparator): The post-operative patients (osteochondral lesion of talus), follow-up with product in live-feedback closed condition.
  After surgery, we will educate the patients about weight bearing protocol on post-op first day and post op 3 week. The protocol is " first 3 weeks, %0 body weight bearing (BWB), second 3 weeks between %10-%20 BWB". Patients' compliance to BWB protocol will be monitored daily with the WBM smart insole system in case live-feedback is turned off. Pre-op and post-op 6 week, we evaluate the patients in case of ankle function, pain with The American Orthopaedic Foot & Ankle Society (AOFAS) Scoring. The relationship with compliance to weight bearing success and AOFAS scores will be evaluate.
  Interventions: Device: With WBM smart insole system to monitor compliance of specified weight bearing limits data in live feedback on and off situations

INTERVENTIONS:
Device: With WBM smart insole system to monitor compliance of specified weight bearing limits data in live feedback on and off situations — Weight Bearing Protocol (Duration: Post-Op. 6 week)
  * Post-op 3 week non-weight bearing (%0 body weight of patient)
  * Post- op 3 week touch down weight bearing (%10-%20 body weight of patient) Group I - monitoring with device while the live feedback mechanism turned on Group II- monitoring with device while the live feedback mechanism turned off

SUMMARY:
Randomized, prospective, double-blind study: Avascular, anöral and non-regenerative cartilage tissue mostly repaired via arthroscopic surgeries. After that, the patients rehabilitate with optimum weight bearing protocols in post-operative and discharge periods by physiotherapists. In the post-operative period, optimum weight bearing is vital for this tissue healing. There is not any opportunity or device to follow up the compliance of patients to weight bearing. We aimed to develop a device with mobile application to monitor the compliance the patients to weight bearing protocols. This device is designed to could give negative live feedback (with visual audible and vibrating warnings) in order to ensure the compliance of patients. Thanks to the device, health professionals will also have the opportunity to monitor the patient's compliance with the protocol on a daily basis. We hypothesized that patients monitored with this device may have a better recovery.

DETAILED DESCRIPTION:
The cartilage tissue, reduces the friction forces in the joints and distributes loads on the joints, is damaged by aging, trauma exposure and degeneration. This tissue is avascular, aneural and non-regenerative. To repair the damaged cartilage tissue arthroplasty method is mostly chosen and the surgery of talus osteochondral lesions is mostly performed type among them. In the post-operative period, optimum weight bearing is vital for this tissue healing. Optimum weight bearing means that the repaired tissue is loaded by a weight which is in between specific percentage of the body weight. During the healing process, educating and compliance of the patients about optimum weight bearing in hospital and after discharge it is difficult to ensure continuity of compliance. At that point the clinical problem arises in terms of teaching the patients the preferred weight bearing percentages (protocols) and their compliance on weight bearing protocols both in hospitalization and home care period. There is not any opportunity or device to follow up the compliance of patients to weight bearing protocols after discharge. A research stated that as the pain symptom decreases, the compliance of patients to optimum weight bearing protocols disappear in home care period even if they had adhered the taught protocol at the clinic. The loss of compliance in the postoperative rehabilitation phase can delay repaired tissue healing and often revision surgery be necessary. This situation necessitated the follow-up of the patients by the physiotherapist using the live-feedback systems. For this purpose, we aimed to develop an android mobile application (system) that will work synchronized with pressure sensors placed under an insole (device). The producing and effectiveness research of mentioned device will consist of two stages. At the first stage will be about product development and testing with volunteer healthy participants. At the second stage named as testing its applicability on patients. The patients will be randomized to two group as Group I (rehabilitate with live-feedback system) and Group II (rehabilitate via system without live- feedback) to evaluate the effectiveness of the live-feedback and mentioned system. The volunteer patients will be evaluated each day, in term of compliance with the weight bearing protocol for 6 weeks. The American Orthopedic Foot Ankle Society, Ankle-hindfoot (AOFAS-AHF) scoring will be administered to each patient on preoperative day and 6 weeks after surgery in order to be evaluate assess the effectiveness of clinical recovery. We expect, thanks to this live feedback system, the health professionals to be capable of determining and monitoring of patients' weight bearing percentages to the body weight during their healing process. Also, the patient will be alerted by the system with visual audible and vibrating warnings, if non-compliance with the weight bearing protocol. Thus, patients can do their own follow-up without a health professional. In this way, continuity of compliance could be ensured. We hypothesized that the development of the insole is expected to help overcome the clinical difficulties encountered during the rehabilitation process and reduce the need for revision operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptomatic osteochondral lesion of the Talus.
* Magnetic resonance of the ankle showing osteochondral injury of a single talus
* People who can use smart phone (andoid or ios)

Exclusion Criteria:

* Recurrent osteochondral lesions of the talus
* Multiple osteochondral lesions
* Severe ankle instability, requiring open repair
* History of a previous foot or ankle surgery of the ipsilateral foot
* Having a systematic disorders like Diabetes Mellitus, Rheumatoid arthritis etc.
* Inability to return to the surgery site to practice long-term follow-up evaluations or lack of readiness to complete the indicated evaluation forms.
* Patients with a qualitative or quantitative commitment that prevents consent or assent their participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Evaluation the clinical recovery of osteochondral lesion of talus post operative patients. | pre-operative day, post-op 6 week, post-op 12 week, post-op 24 week
  American Orthopedic Foot and Ankle Society- Ankle hindfoot scale will be used for this evaluation. The scale includes nine items that can be divided into three sub-scales (pain, function and alignment). Pain consists of one item with a maximal score of 40 points, indicating no pain. Function consists of seven items with a maximal score of 50 points, indicating full function. Alignment consists of one item with a maximal score of 10 points, indicating good alignment. The maximal score is 100 points, indicating no symptoms or impairments. This scale will be used for evaluation the clinical recovery of osteochondral lesion of talus post operative patients.

OTHER OUTCOMES:
Monitoring the compliance with weight bearing protocol | Post-op every day for 6 weeks
  number of times above the specified upper threshold, the number of failures to reach the specified lower threshold, percentage of steps in correct weight bearing range parameter will be monitored by the device (insole with pressure sensors)
Visual Analog Scale | Post-op every day for 6 weeks, post-op 12 week, post-op 24 week
  Visual Analog Scale for Pain (VAS-Pain): a pain rating scale based on self-reported measures of symptoms. A 10cm line numbered from 0 to 10 represents a continuum between "no pain" (zero) and "worst pain" (ten). It can also be interpreted as a 0-to-100 points score.
  This scale will be used for assessment of patient's pain levels after activity and at rest

CONTACTS AND LOCATIONS:
Overall Officials: İlkşan Demirbüken, Assoc.Prof., Study Chair — Marmara University; Ender Ersin AVCI, MsC, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No